CLINICAL TRIAL: NCT02274805
Title: Collection of Human Tissue Samples From the Neck Region for Characterization of Its Molecular and Biochemical Signatures
Acronym: Human BAT
Status: Active, not recruiting | Type: Observational
Sponsor: AdventHealth Translational Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: TRIMD FH 644456
Record Dates: First submitted 2014-09-09; First posted 2014-10-24 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Obesity
Keywords: Brown adipose tissue; Neck surgery
MeSH Terms: conditions — Obesity | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Muscle and adipose tissue from the neck region, and blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Adults presenting for surgery in the neck area
  Interventions: Procedure: Adults presenting for surgery in the neck area

INTERVENTIONS:
Procedure: Adults presenting for surgery in the neck area

SUMMARY:
The purpose of the study is to gather tissue (from the neck region), specimens (blood and urine) and medical record data from many patients and store them in one place so that scientists have the information they need to conduct research and learn about new ways to predict, identify and treat illness, specifically those related to obesity and diabetes.

DETAILED DESCRIPTION:
This protocol is designed to actively collect biospecimens (specifically, tissue from the neck region) and clinical data for donation to the TRI-MD, specifically, Dr. Sparks' laboratory. These specimens and data will be available to Dr. Sparks for future research activity in accordance with the Florida Hospital and Translational Research Institute for Metabolism and Diabetes (TRI) policies.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 and older presenting for surgery in the neck area
* Able to provide informed consent

Exclusion Criteria:

* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a protocol for the collection of muscle and adipose tissues from patients of Dr. Alric Simmonds undergoing surgery in the neck region as part of their clinical care. In addition to the tissues collected at the time of the procedure, these patients will also be asked to provide additional blood samples before their procedure either at their pre-operative visit or on the morning of the surgery.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2014-11; Primary Completion 2019-04-25 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Collection of brown adipose neck tissue | Day of scheduled surgery
  Any tissue deemed suitable by the surgeon and/or the research team during the neck surgery for the study's research objectives will be removed and collected for donation to this protocol. When there is enough tissue available, half will be snap frozen for extraction of DNA, RNA and protein. The other half will be cryopreserved for the future production of viable cells. When there is not enough tissue, the person collecting the samples will determine the processing. For research purposes, we aim to collect up to 500mg of each tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Sparks, PhD, Principal Investigator — Translational Research Institute for Metabolism and Diabetes
Locations (1):
- Translational Research Institute for Metabolism and Diabetes, Orlando, Florida, United States

REFERENCES:
- [Background] van Marken Lichtenbelt WD, Vanhommerig JW, Smulders NM, Drossaerts JM, Kemerink GJ, Bouvy ND, Schrauwen P, Teule GJ. Cold-activated brown adipose tissue in healthy men. N Engl J Med. 2009 Apr 9;360(15):1500-8. doi: 10.1056/NEJMoa0808718. PMID 19357405
- [Background] Cypess AM, Lehman S, Williams G, Tal I, Rodman D, Goldfine AB, Kuo FC, Palmer EL, Tseng YH, Doria A, Kolodny GM, Kahn CR. Identification and importance of brown adipose tissue in adult humans. N Engl J Med. 2009 Apr 9;360(15):1509-17. doi: 10.1056/NEJMoa0810780. PMID 19357406
- [Background] Wijers SL, Schrauwen P, Saris WH, van Marken Lichtenbelt WD. Human skeletal muscle mitochondrial uncoupling is associated with cold induced adaptive thermogenesis. PLoS One. 2008 Mar 12;3(3):e1777. doi: 10.1371/journal.pone.0001777. PMID 18335051
- [Background] Vijgen G, van Marken Lichtenbelt W. Brown adipose tissue: clinical impact of a re-discovered thermogenic organ. Front Biosci (Elite Ed). 2013 Jun 1;5(3):823-33. doi: 10.2741/e663. PMID 23747899
- [Background] Vijgen GH, Bouvy ND, Leenen L, Rijkers K, Cornips E, Majoie M, Brans B, van Marken Lichtenbelt WD. Vagus nerve stimulation increases energy expenditure: relation to brown adipose tissue activity. PLoS One. 2013 Oct 23;8(10):e77221. doi: 10.1371/journal.pone.0077221. eCollection 2013. PMID 24194874
- [Background] Vijgen GH, Sparks LM, Bouvy ND, Schaart G, Hoeks J, van Marken Lichtenbelt WD, Schrauwen P. Increased oxygen consumption in human adipose tissue from the "brown adipose tissue" region. J Clin Endocrinol Metab. 2013 Jul;98(7):E1230-4. doi: 10.1210/jc.2013-1348. Epub 2013 Jun 19. PMID 23783102
- [Background] van der Lans AA, Hoeks J, Brans B, Vijgen GH, Visser MG, Vosselman MJ, Hansen J, Jorgensen JA, Wu J, Mottaghy FM, Schrauwen P, van Marken Lichtenbelt WD. Cold acclimation recruits human brown fat and increases nonshivering thermogenesis. J Clin Invest. 2013 Aug;123(8):3395-403. doi: 10.1172/JCI68993. Epub 2013 Jul 15. PMID 23867626
- [Background] Vosselman MJ, Brans B, van der Lans AA, Wierts R, van Baak MA, Mottaghy FM, Schrauwen P, van Marken Lichtenbelt WD. Brown adipose tissue activity after a high-calorie meal in humans. Am J Clin Nutr. 2013 Jul;98(1):57-64. doi: 10.3945/ajcn.113.059022. Epub 2013 May 29. PMID 23719558
- [Background] van Rooijen BD, van der Lans AA, Brans B, Wildberger JE, Mottaghy FM, Schrauwen P, Backes WH, van Marken Lichtenbelt WD. Imaging cold-activated brown adipose tissue using dynamic T2*-weighted magnetic resonance imaging and 2-deoxy-2-[18F]fluoro-D-glucose positron emission tomography. Invest Radiol. 2013 Oct;48(10):708-14. doi: 10.1097/RLI.0b013e31829363b8. PMID 23695084
- See also: Florida Hospital Translational Research Institute for Metabolism and Diabetes — http://www.tri-md.org